CLINICAL TRIAL: NCT02061943
Title: Validity and Reliability of the Spasmodic Dysphonia Diagnosis and Assessment Procedure (SD-DAP) for Quantifying Symptom Change
Brief Title: Examining the Spasmodic Dysphonia Diagnosis and Assessment Procedure (SD-DAP) for Measuring Symptom Change
Status: Withdrawn | Type: Observational
Why Stopped: Study not started
Sponsor: Emory University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Office of Rare Diseases (ORD) (NIH)
Responsible Party: Principal Investigator, Hyder A. Jinnah, MD, PhD, Principal Investigator, Emory University
Other Study IDs: IRB00068259; U54NS065701 (NIH)
Record Dates: First submitted 2014-02-11; First posted 2014-02-13 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Spasmodic Dysphonia; Laryngeal Dystonia
Keywords: Spasmodic dysphonia; Laryngeal dystonia; Dystonia; Severity
MeSH Terms: conditions — Dysphonia; Dystonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a study of patients with spasmodic dysphonia to determine how best to measure the severity of the disorder in patients. It addresses which characteristics of speech are the best indicator of whether or not a particular treatment has benefited a person with spasmodic dysphonia. We hope to recruit 20 participants each at 2 different centers. The evaluation for each participant will be done on a two visits, one just before and another several weeks after treatment.

DETAILED DESCRIPTION:
This is a study of changes in voice and laryngeal function with treatment recorded using the Spasmodic Dysphonia Diagnosis and Assessment Procedure (SD-DAP). Persons with adductor spasmodic dysphonia will complete a questionnaire on the Voice Handicap Index (VHI) and ratings of speech effort as well as have their speech recorded and receive a nasolaryngoscopy examination prior to their usual treatment with botulinum toxin injection into the laryngeal muscles for their voice disorder. They will return for re-examination several weeks later after their injection and repeat each of the examinations. The purpose is to determine which items on the SD-DAP are sensitive to changes in the severity of their voice disorder. The items that show sensitivity would be those that would be useful for assessing voice outcomes in clinical trials. Some of the questions this study is trying to answer are

* What is the best way to measure the severity of spasmodic dysphonia?
* How does treatment of spasmodic dysphonia by botulinum toxin injection affect voice for communication in regular daily life in spasmodic dysphonia
* Is change in speaking effort related to the change in severity of spasmodic dysphonia with botulinum toxin injection?

Each participant in this study will be asked to do the following:

* Provide a copy of medical records and medical history relating to the diagnosis of spasmodic dysphonia.
* Have an examination by an otolaryngologist with a medical periscope inserted in the throat to view the voice box in action. The examination will be so it can be reviewed later by several different experts.
* Complete questionnaires regarding the severity of their disorder before and after receiving their usual treatment; an injection of botulinum toxin into the laryngeal muscles.
* Repeat a speech recording and laryngeal examination before and after treatment

ELIGIBILITY:
Inclusion Criteria:

* be clinically diagnosed with primary spasmodic dysphonia (laryngeal dystonia)
* be 18 years of age or older

Exclusion Criteria:

* be diagnosed with secondary spasmodic dysphonia (laryngeal dystonia)
* be younger than 18 years of age
* unable to complete questionnaires
* not able to have a nasolaryngoscopy (examination of the voice box with a medical periscope)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with spasmodic dysphonia are eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
SD-DAP | 2-4 weeks
  Identify items within the SD-DAP that are sensitive to symptom reduction when participants with spasmodic dysphonia are treated with botulinum toxin.

CONTACTS AND LOCATIONS:
Overall Officials: Christy Ludlow, PhD, Principal Investigator — James Madison University
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Washington University in St. Louis, St Louis, Missouri